CLINICAL TRIAL: NCT06806254
Title: Attitude and Practice for Deep Caries Management Between Egyptian and Indian Dentists. a Cross -Sectional Study
Brief Title: Attitude and Practice for Deep Caries Management Between Egyptian and Indian Dentists : a Cross Sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fahme Liyakath pk, Principle investigator, Cairo University
Other Study IDs: Deep Caries Cross section
Record Dates: First submitted 2025-01-05; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Deep Dental Caries
Keywords: Deep Caries; Dentine caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Study type: Observational Study To assess and compare the attitudes, and practices of dentists in Egypt and India regarding the removal of deep dentin caries and preferred restorative strategies. In addition to correlate between dentist's understanding of caries and its treatment and factors such as age, gender, degree of education and clinical setting.

DETAILED DESCRIPTION:
Study type:Observational study To evaluate and compare the views and practices of dentists in Egypt and India concerning the removal of deep dentin caries and their preferred restorative approaches. Additionally, the study aims to examine the relationship between dentists' understanding of caries and its treatment, along with factors such as age, gender, level of education, and clinical environment.

primary outcome-Attitudes, and practices of dentists in Egypt and India regarding the removal of deep dentin caries and their preferred restorative strategies.

secondary outcome:The relationship between dentists' attitudes and their practices in managing deep caries treatment may be affected by factors such as age, gender, education level, and clinical experience.

comparison groups: Population (P1): Dentists practicing in Egypt

- Population(P2) : Dentists practicing in India

ELIGIBILITY:
Inclusion Criteria:

* Inclusion: Licensed dentists actively practicing in Egypt or India.

Exclusion Criteria:

* Exclusion: Dentists not currently practicing or recent graduates without practical experience

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dentists (at various levels of education and years of practice) practicing in Egypt and India: Educational Background: Various qualifications, such as dental degrees and specialized training. Years of Practice: Categories of experience: less than 5 years, 5-10 years, and over 10 years. Geographic Location: Dentists from diverse urban and rural regions.
Sampling Method: Non-Probability Sample
Enrollment: 766 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Attitude of practicing patient in Egypt and India regarding deep caries management | Through study completion,an average of 3 months
  Current Attitude and how dentist think regarding strategies of deep caries management either complete caries removal or partial/ selective caries removal. And which is thought to be the most rationalized concept to use according to each dentist. This will be done using a previously validated questionaire

SECONDARY OUTCOMES:
Practice of Egyptian and Indian dentist to deep caries management practices | Through study completion,an average of 3 months
  The adopted strategy the dentist practices in daily management of deep caries lesions. This will be measured using a previously validated questionnaire
Impact of demographic data on dentist attitude and practice regarding deep caries management | Through study completion,an average of 3 months
  Impact of each of age, gender, geographic location , educational level and experience of dentists on how they think about caries management strategies and how they practice it.
  Each variant will be analyzed statistically solely. Demographic data will be collected by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Iman El Sayad, Iman El Sayad, Study Director — Professor of Conservative Dentistry, Faculty of Dentistry Cairo University
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided